CLINICAL TRIAL: NCT06255405
Title: The Effects of Dyadic Parent-child Self-compassion Program on Children' Psychological Well-being: A Pilot Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Metropolitan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HE-SF2022/03
Record Dates: First submitted 2024-02-04; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Psychological Well-Being
Keywords: psychological well-being; self-compassion; children
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Intervention group (Experimental): Dyadic parent-child self-compassion program will be provided.
  Interventions: Behavioral: Self-compassion
- Waitlist control group (No Intervention): Participants in the control group will be instructed to live their lives as usual, no intervention will be imposed during study period. They will be provided with the program after the study.

INTERVENTIONS:
Behavioral: Self-compassion — The dyadic parent-child self-compassion program is designed by the research team and validated by a panel of experts. It includes 5 weekly sessions. Each session lasts for 60 minutes. The dyads will be guided to do self-compassion practices (e.g. affectionate breathing, compassionate letters to oneself etc). Didactic topics, inquiry, and home practices are also involved.
  Arms: Experimental: Intervention group

SUMMARY:
Suboptimal psychological well-being in children can have substantial negative effects on their physical health, academic performance, and lifelong health. Preliminary evidence supports that self-compassion have positive impacts on psychological well-being in elderly, adults, and adolescents, but there is apparently lack of this kind of evidence in children. Involvement of parents in the program potentially optimize the effects, this study thus designs a dyadic parent-child self-compassion program (DPC-SC) and aim to examine its effects on children's psychological well-being.

ELIGIBILITY:
Inclusion Criteria: (Child)

* Study in Primary three or four.
* Can communicate in Cantonese.

Exclusion Criteria: (Child)

* Have emotional dysregulation
* Have past history of mental illness
* Recently experience trauma
* Are in an acute health crisis

Inclusion Criteria: (Parents)

* Is the primary caretaker of the children
* Is willing to interact and do the practices with their children
* Can communicate in Cantonese
* Commit to attend all sessions

Exclusion Criteria: (Parents)

* Have emotional dysregulation
* Have past history of mental illness
* Recently experience trauma
* Are in an acute health crisis

Ages: 8 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Psychological well-being (child) | Baseline, immediately after intervention
  Chinese version of the Psychological Well-Being Scale (C-PWBS)

SECONDARY OUTCOMES:
Perceived stress levels (Child) | Baseline, immediately after intervention
  Chinese version of the 10-item Perceived Stress Scale (PSS-10)
Self-compassion levels (Child) | Baseline, immediately after intervention
  Chinese version of the Self-Compassion Scale for Youth (SCS-Y)
Self-compassion levels (parents) | Baseline, immediately after intervention
  Chinese version of the self-compassion scale (SCS)

CONTACTS AND LOCATIONS:
Overall Officials: Wai Man Sin, MN, Principal Investigator — Hong Kong Metropolitan University